CLINICAL TRIAL: NCT05462951
Title: Phase 0 Clinical Trial of Molecular Biomarkers in Women With Uterine Cervix Cancer
Brief Title: Clinical Trial of Molecular Biomarkers in Women With Uterine Cervix Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Denise Fabian (Other)
Collaborators: UK Radiopharma Alliance (Unknown)
Responsible Party: Sponsor-Investigator, Denise Fabian, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: MCC-22-GYN-09
Record Dates: First submitted 2022-07-08; First posted 2022-07-18 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Uterine Cervix Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Radiochemotherapy followed by brachytherapy: Standard daily radiotherapy plus weekly cisplatin followed by brachytherapy
  Interventions: Radiation: Standard

INTERVENTIONS:
Radiation: Standard — Radiation then brachytherapy

SUMMARY:
This is a phase 0 clinical trial of molecular biomarkers in women with uterine cervix cancer. Women receive standard-of-care radiochemotherapy followed by brachytherapy. Blood samples are obtained to detect circulating levels of deoxyribonucleotides, human papillomavirus DNA, and circulating tumor cells.

ELIGIBILITY:
Inclusion Criteria:

- Untreated pathologically or cytologically-confirmed diagnosis of stage IB3 (> 4cm), II, III, or IVA (FIGO 2018) squamous, adenosquamous, or adenocarcinoma of the uterine cervix not amenable to curative surgery alone.

Exclusion Criteria:

* Presence of another concurrent active invasive malignancy
* Prior invasive malignancy diagnosed within the last three years except for [1] non-melanoma skin cancer or [2] prior in situ carcinoma of the cervix
* prior pelvic radiotherapy for any reason that would contribute radiation dose that would exceed tolerance of normal tissues at the discretion of the treating physician.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an unblinded phase 0 window-of-opportunity intervention clinical trial to study biomarkers of uterine cervix cancer biology and disease progression in women undergoing cisplatin-based radiochemotherapy for advanced-stage uterine cervix cancer.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Biomarker | 3 months posttherapy
  deoxyribonucleotide levels
Biomarker | 3 months posttherapy
  HPV DNA levels
Biomarker | 3 months posttherapy
  Circulating tumor cell count

CONTACTS AND LOCATIONS:
Overall Officials: Denise Fabian, MD, Principal Investigator — University of Kentucky
Locations (1):
- Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No